CLINICAL TRIAL: NCT07026734
Title: Effects of Deep Brain Stimulation (DBS) on Laryngeal Function and Associated Behaviors in Parkinson Disease
Brief Title: The Impact of Deep Brain Stimulation on Speech and Swallow Function in Parkinson Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB202300382; R01DC020450 (NIH)
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Parkinson disease; Deep brain stimulation; voice; speech; swallow
MeSH Terms: conditions — Parkinson Disease; Speech

STUDY DESIGN:
Intervention Model Description: The "intervention" is deep brain stimulation, and this is being done in the context of routine clinical care (i.e., the participants are not allocated to the GPi or STN by the study; this decision is made by the clinical team). The study investigates the pre/post DBS impact on laryngeal function and other laryngeal mediated behaviors, such as voice, swallow, and cough.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPi DBS (Other): People with PD who are approved to receive deep brain stimulation (DBS) surgery to the globus pallidus internal segment.
  Interventions: Procedure: Deep brain stimulation surgery - GPi
- STN DBS (Other): People with PD who are approved to receive deep brain stimulation (DBS) surgery to the subthalamic nucleus.
  Interventions: Procedure: Deep Brain Stimulation Surgery - STN

INTERVENTIONS:
Procedure: Deep brain stimulation surgery - GPi — Deep brain stimulation (DBS) surgery will be performed as normal clinical care. People with PD who are approved for GPi DBS will be enrolled in the study prior to their surgery.
  Arms: GPi DBS
Procedure: Deep Brain Stimulation Surgery - STN — Deep brain stimulation (DBS) surgery will be performed as normal clinical care. People with PD who are approved for STN DBS will be enrolled in the study prior to their surgery.
  Arms: STN DBS

SUMMARY:
Nearly one-million people in North America are now living with Parkinson's disease (PD), and that number is projected to rise to nearly 1.2 million by 2030. With advancements in neuromodulatory technologies, increasingly more of these individuals elect to undergo deep brain stimulation (DBS) surgery in order to control symptoms of the disease, including refractory tremor, medication-induced dyskinesias, and PD-associated dystonia. The two most common DBS neural targets for controlling these symptoms are the globus pallidus internal segment (GPi) and the subthalamic nucleus (STN). Recent meta-analyses have shown relative equivalence between these two sites at controlling core PD symptoms. To date, there is not conclusive evidence regarding the potential impact of DBS to GPi or STN on laryngeal-mediated functions of voice, swallowing, and cough, and consequently no guidance on whether these outcomes should be considered when selecting DBS target. Therefore, the goal of this project is to determine the impact of DBS neural target (STN versus GPi), lead location within the target, laterality, and stimulation settings on voice, swallow and cough function in people with PD. The larynx is an important player in each of these functions, and our central hypothesis is that spread of stimulation to corticobulbar fibers in the genu of the internal capsule have deleterious effects on laryngeal motor control, resulting in voice, swallow, and cough dysfunction. We have identified three specific aims for this application: 1.) To compare laryngeal function during volitional voice tasks pre-post DBS, and when DBS placement is bilateral versus unilateral for STN and GPi targets. 2.) To compare laryngeal function during volitional and induced cough tasks pre-post DBS, and when DBS placement is bilateral versus unilateral for STN and GPi targets. 3.) To compare airway safety associated with laryngeal onset, degree, and duration of maximum closure during swallowing, pre-post DBS, and when DBS placement is bilateral versus unilateral for STN and GPi targets. These hypotheses were developed based on compelling published and unpublished preliminary data. We will accomplish these aims by enrolling people with PD who are being considered for DBS surgery. We will measure physiologic, functional, and quality of life parameters of voice, swallow and cough pre- and post-surgically. The realization of the proposed aims is significant because it will address a substantial gap in our understanding of DBS outcomes related to communication and airway protection, which are important in terms of morbidity, mortality, and quality of life for patients with PD. The translational potential to provide additional guidance to DBS surgical teams regarding whether voice, swallow or cough functions should be considered with selecting DBS target and/or laterality is high. Ultimately, the project fits squarely within the overarching goal of the research team to deliver the best possible care to people with PD.

DETAILED DESCRIPTION:
Parkinson disease (PD) is among the most common neurodegenerative conditions affecting adults worldwide, with estimated prevalence in the United States to reach 1.2 million by the year 2030. In addition to the hallmark motor symptoms of PD, people with PD also experience changes to functions of communication and airway protection, in particular deficits in voice production, swallowing, and cough, and these contribute considerably to the morbidity and mortality of PD. Deep Brain Stimulation (DBS) is an increasingly used therapeutic option for alleviating many of the motor symptoms of PD; however, the impact of DBS on voice, swallowing, and cough is not clear. DBS targeted nuclei for PD include the subthalamic nucleus (STN) and globus pallidus interna (GPi). While historical reports suggested different therapeutic effectiveness for limb motor outcome across DBS target sites, more recent data suggest equipoise in treatment outcomes for STN and GPi targets. There is less conclusive evidence on the impact of DBS target site or laterality on voice, swallow, or cough, with existing evidence largely limited to bilateral STN DBS outcomes. Further, of the extant literature, interpretation of outcomes is limited by the methods employed that may lack longitudinal objective and validated outcomes pre- and post- DBS surgery, ON and OFF DBS stimulation, or that incorporate neurostimulation parameters or functional connectivity to adjacent brain regions in their design. Thus, although DBS is now routinely used in PD, significant gaps in knowledge remain regarding the impact of this therapeutic adjuvant on communication and airway protection.

The current project proposes to evaluate the effects of STN or GPi DBS placement for treating limb symptomatology, on voice, cough, and swallowing functions. We hypothesize that DBS stimulation at these sites will impact laryngeal motor control affecting voice, cough, and swallow functions due to spread of stimulation to cortibobulbar pathways. Because cranial nerve nuclei receive predominately bilateral upper motor neuron innervation, we posit that DBS effects are exacerbated with bilateral placement and stimulation of either the STN or GPi sites. Evidence that bilateral lesional stereotactic surgeries such as pallidotomy, capsulotomy and/or thalamotomy lead to worsening bulbar function, are in line with this hypothesis. Our supporting preliminary DBS data indicate that metrics of voice and swallowing degrade significantly following DBS to either the STN or GPi target, however measures of cough effectiveness may actually improve. Our innovative, multidisciplinary approach to determining DBS candidacy, target, and laterality provides an ideal opportunity to prospectively study these outcomes in a rigorous, pragmatic and methodical way. Therefore, we seek to address the following specific aims:

1. To compare laryngeal function during volitional voice tasks pre-post DBS, and when DBS placement is bilateral versus unilateral for STN and GPi targets. Hypothesis 1a: Laryngeal function during volitional voice tasks will remain unchanged pre-post unilateral STN or GPi DBS targets. Hypothesis 1b: Laryngeal function during volitional voice tasks will be worsened pre-post bilateral STN or GPi DBS.
2. To compare laryngeal function during volitional and induced cough tasks pre-post DBS, and when DBS placement is bilateral versus unilateral for STN and GPi targets. Hypothesis 2a: Peak expiratory cough airflow and cough volume acceleration will not significantly change for either voluntary or induced cough pre-post unilateral DBS placement to the STN and GPi targets. Hypothesis 2b: Peak expiratory cough airflow and volume acceleration will be increased during volitional cough compared to induced cough in those with bilateral DBS placement to the STN and GPi targets compared to pre-DBS.
3. To compare airway safety associated with laryngeal onset, degree, and duration of maximum closure during swallowing, pre-post DBS, and when DBS placement is bilateral versus unilateral for STN and GPi targets. Hypothesis 1: Swallowing safety, along with the degree, and duration of maximum laryngeal vestibule closure (LCV) during videofluoroscopic evaluation will be significantly reduced pre-post bilateral DBS placement to the STN and GPi targets compared to unilateral STN and GPi DBS treatment.

This prospective clinical trial will include two participant groups: STN DBS group and GPi DBS group. Each group will complete 4 study visits spaced approximately 6 - 12 months apart. For both the STN and GPi DBS groups, the first study visit will be completed following approval for surgery, but prior to DBS surgery. The second visit will follow placement of their first (unilateral) DBS lead, lead activation, and programming, and the third visit will follow placement of the second (bilateral) lead, lead activation, and programming (see Figure 1 for surgical timeline at our institution). The 4th visit will occur 6 - 12 months following the third visit to account for any time-related changes that may occur following DBS. The post-surgical visits will be completed across two days: one with the stimulators on, and the other with them off. The rationale for including stimulator on / off conditions relates to the central hypothesis: we hypothesize that spread of stimulation to corticobulbar fibers leads to changes in laryngeal motor control; therefore, we expect measures made in the off-stimulation condition NOT to differ from the pre-surgical baseline measures. For stimulation-off condition, participants will arrive for their appointment having turned off the stimulators overnight, which is standard care for their DBS follow-up visits. In order to maintain a reasonably low level of participant burden, all study assessments will be completed with participants in the medication 'on' state. However, we will collect data from their DBS programming visits which do assess patients in an off-medication state to document medication-related motor outcomes.

In order to complete this project in a pragmatic fashion that respects the best medical management for participants, we will not randomize participants to receive/not receive DBS, or to DBS target. DBS to both the STN and GPi has been FDA approved for use to treat motor features of PD since 2002; it will be used in a manner consistent with the population and indication for which it was approved. The DBS groups will consist of people who are already approved for DBS surgery (i.e., they are NOT receiving DBS because of participation in this study), and the control group will be recruited from over 1700 people with PD currently followed prospectively in our IRB-approved database, who do not have existing DBS and are not currently being considered for DBS. The DBS target site will be determined in the usual manner by the clinical DBS team based on factors such as motor concerns or complications, cognitive status and individual goals of the surgery, as per guidance by the Congress of Neurological Surgeons. Our inclusion criteria specifies that only patients with mild, or moderate voice and swallowing function may participate. Our goal with this approach is to increase the likelihood of well-matched GPi versus STN groups in terms of their pre-surgical voice and swallow functions, but not to interfere with surgical decisions and standard patient care.

Procedures Participant demographics: Demographic information, including age, sex, disease duration, primary goals for DBS surgery, stimulation parameters and levodopa equivalent dose.

Motor outcomes: Because DBS is intended to alleviate the motor symptoms of PD, it will be important to assess whether this primary therapeutic goal is achieved. Specifically, we will record:

* Unified Parkinson's Disease Rating Scale, Hoehn (UPDRS) - Will be used to assess change in motor function of participants. This will be collected both on/off medication and on/off stimulation.
* Hoehn & Yahr score - To monitor disease stage. Pulmonary function measures: In order to account for physiologic changes in the respiratory system as possible contributing factors, we will analyze pulmonary function in all participants. The forced expired volume in the first second (FEV1) of a forced vital capacity (FVC) maneuver will be measured for each participant using a digital spirometer (Spirovision 3+m, Futuremed; or Koko spirometry, Nspire health). Maximum inspiratory pressure (PiMax) and maximum expiratory pressure (PeMax) will be measured with a manometer (MicroRPM, Micromedical inc). We will use standard procedures, as put forth by the American Thoracic Society, for measuring FVC, FEV1, the ratio of FEV1/FVC, PiMax, and PeMax.

Cognition: There is known impact of DBS and/or PD disease progression on cognitive function 15,50. In order to first screen for the presence of moderate or severe cognitive impairment (part of exclusionary criteria), as well as to account for potential impact cognitive changes on task performance, the Montreal Cognitive Assessment (MoCA) will be administered by a researcher trained and certified to administer the test (per most recent guidelines for administration on mocatest.org). This will be performed at each study visit.

Laryngeal imaging procedures: Indirect laryngoscopy will be performed with a flexible endoscope. Participants will be seated in a dental exam chair in the upright position. Water-based lubricant will be used to coat the endoscope which will be passed trans-nasally. Once the endoscope is in place with the larynx and surrounding structures clearly visible, the participant will be asked to perform the following tasks, three times each: rest breathing, breath hold, laryngeal diadochokinesis (alternating /i/ and brisk sniff), sustained vowel phonation, pitch glides up and down, soft voluntary cough production, and counting from sixty to seventy, and from eighty to ninety. Participants will be instructed to perform these tasks at normal pitch and loudness levels

Audio-perceptual & Acoustic Procedures: Participant speech samples will be collected in a quiet clinical research space. Participants will be fitted with a head-mounted microphone situated 10 cm and 45° to 50° angle from the corner of the mouth54,55. Participants will also be equipped with electroglottography (EGG) sensors that are placed on the lateral aspects of the neck, on either side of the thyroid notch (Glottal Enterprises EG2-PCX2). The electrodes are held in place by a strap that is placed around the neck and secured with Velcro. Electrode gel may be used to improve the signal fidelity. They will perform various speech tasks.

Voluntary Cough: Participants will be outfitted with a facemask covering the nose and mouth. The facemask will be coupled to a pneumotachograph and differential pressure transducer. The cough airflow signal will be digitized (Power Lab Data Acquisition System) and recorded (LabChart 7; ADInstruments, Inc) to a laptop computer. Participants will be asked to cough 3 times, with the instruction to "cough as if something went down the wrong pipe.

Induced Cough: Participants will be outfitted with the same equipment used for voluntary cough testing, however there will be a side port with a one-way inspiratory valve for nebulizer connection. The nebulizer will be connected to a dosimeter that delivers aerosolized capsaicin solution during inspiration with a delivery duration of 2 seconds. Participants will complete a capsaicin challenge with three randomized blocks of 0, 50, 100, 200, and 500 μM capsaicin dissolved in a vehicle solution. Participants will be given the instruction "cough if you need to" prior to capsaicin delivery.

Swallowing Evaluation: Swallowing function and physiology will be assessed using high resolution digital fluoroscopy at a pulse rate of 30 frames per second, digitally stored for retrieval and offline analysis. Participants will be seated in the lateral viewing plane. Participants will perform trials thin and pudding-thick boluses.

These tasks will be performed at each study visit, and in the on/off DBS conditions post surgically.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of idiopathic (non-genetic/familial) PD made by fellowship-trained neurologist by applying strict UK brain bank criteria

Hoehn & Yahr staging I - IV

Approved for DBS surgery to either STN or GPi, with NO existing DBS electrodes.

Mild or moderate voice / swallow problems

Exclusion Criteria:

Neurological disorder(s) other than PD (including essential tremor) Severe neuropsychological dysfunction, unstable psychiatric disease at the discretion of the treating neurologist/psychiatrist (i.e., severe depression) or moderate to severe cognitive impairment.

History of:

* Head, neck, or lung cancer (except minor squamous cell skin cancers)
* Structural, functional, or neurologic voice disorder unrelated to PD
* Chronic refractory cough
* Bleeding disorder

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Glottal closure | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  Flexible or rigid endoscopy will be used to image the larynx. From these images, glottal closure will be analyzed using a 6-point scale ranging from 1 (complete glottal closure along all length of the vocal folds) and 6 (Incomplete glottal closure along all length of the vocal folds)
Voluntary cough airflow | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  The airflow signal from the voluntary cough task will be measured to determine peak airflow, total volume of airflow, and rise time to peak flow.
Swallowing safety | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  The penetration-aspiration scale will be used to determine whether swallowed material enters the airway, and how far down it goes (i.e., above, at, or below the level of the vocal folds) and whether there is visible residue.

SECONDARY OUTCOMES:
Normalized glottal gap area | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  Flexible or rigid endoscopy will be used to image the larynx. From these images, the normalized glottal gap area will be measured. This will be computed by measuring the length of the vocal fold (pixels) and the area of maximum closure achieved during phonation.
Acoustic voice analysis | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  Based on the voice and speech tasks participants perform, praat will be used to analyze the acoust properties of the sound signals.
Audio-perceptual analysis | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  The CAPE-V will be used to analyze the voice and speech tasks by an expert audio-perceptual rater.
EGG | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  Electroglottography will be used to analyze the open quotient based on the vowel prolongation tasks.
Patient reported outcome - VHI | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  Participants will complete the voice handicap index (VHI), which is a 30-item scale asking questions pertaining to how the voice affects various aspect of life.
Induced cough airflow | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  The airflow signal from the induced cough task will be measured to determine peak airflow, total volume of airflow, and rise time to peak flow.
Induced cough sensitivity | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  After each induced cough task, participants are asked to rate their urge to cough on a modified borg scale. The rating of urge to cough serves as a measure of perceived cough sensitivity.
Patient reported outcome - EAT 10 | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  Participants will fill out the EAT-10, which is a self-administered 10-item questionnaire developed to evaluate patients' self-perceived symptoms of swallowing problems.
Swallow timing | Prior to DBS surgery, 4 - 12 months following DBS surgery, and 6 - 12 months after the last post-operative visit
  Based on the imaged swallow, the time of swallow events including onset of pharyngeal phase and duration of laryngeal vestibule closure, will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hegland, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No